CLINICAL TRIAL: NCT00600535
Title: A Pharmacokinetics Study to Assess the Oral Administration of CB7630 (Abiraterone Acetate) Capsule Formulation and Tablet Formulation in Patients With Prostate Cancer
Brief Title: A Pharmacokinetics Study to Assess Abiraterone Acetate Capsule and Tablet Formulations in Patients With Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cougar Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR016933; COU-AA-BE (Other: Cougar Biotechnology)
Record Dates: First submitted 2008-01-14; First posted 2008-01-25 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-04

CONDITIONS: Prostate Neoplasms
Keywords: Prostate neoplasms; Abiraterone acetate; CB7630; Prostate cancer; Pharmacokinetics
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Abiraterone acetate (non-fasting) (Experimental)
  Interventions: Drug: Stage 1 Group 1: abiraterone acetate; Drug: Stage 1 Group 2: abiraterone acetate; Drug: Stage 2: abiraterone acetate
- Abiraterone acetate (fasting) (Experimental)
  Interventions: Drug: Stage 1 Group 1: abiraterone acetate; Drug: Stage 1 Group 2: abiraterone acetate; Drug: Stage 2: abiraterone acetate; Drug: Stage 3: abiraterone acetate; Drug: Stage 3: glucocorticoid; Drug: Stage 4: abiraterone acetate; Drug: Stage 4: glucocorticoid

INTERVENTIONS:
Drug: Stage 1 Group 1: abiraterone acetate — 1000 mg capsules/day orally on Day 1. On Day 8, patients will crossover and receive tablet formulation at the same dose.
Drug: Stage 1 Group 2: abiraterone acetate — 1000 mg tablets/day orally on Day 1. On Day 8, patients will crossover and receive capsule formulation at the same dose.
Drug: Stage 2: abiraterone acetate — 1000 mg tablets/day orally for 12 cycles (28 days/cycle) according to assigned group from Stage 1.
Drug: Stage 3: abiraterone acetate — 1000 mg tablets/day orally for 12 cycles (28 days/cycle).
  Arms: Abiraterone acetate (fasting)
Drug: Stage 3: glucocorticoid — prednisone/prednisolone 5 mg twice daily orally or dexamethasone 0.5 mg once daily for 12 cycles (28 days/cycle).
  Arms: Abiraterone acetate (fasting)
Drug: Stage 4: abiraterone acetate — 1000 mg tablets/day orally for up to 24 cycles (28 days/cycle).
  Arms: Abiraterone acetate (fasting)
Drug: Stage 4: glucocorticoid — prednisone/prednisolone 5 mg twice daily orally or dexamethasone 0.5 mg once daily for up to 24 cycles (28 days/cycle).
  Arms: Abiraterone acetate (fasting)

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics (how the drug concentrations change over time) of capsule and tablet formulations of CB7630 (abiraterone acetate) taken with and without food in patients with prostate cancer.

DETAILED DESCRIPTION:
This is an open-label study (identity of assigned study drug will be known) to evaluate the pharmacokinetics of abiraterone acetate in patients with prostate cancer. The study will be conducted in 4 stages: Stage 1 will measure blood levels after patients take 1 daily dose of abiraterone tablet or capsule formulations with and without food; Stage 2 will measure blood levels of single daily doses of abiraterone tablet formulation taken with or without food in parallel design until disease progression (up to 12 cycles [28 days per cycle]); Stages 3 and 4 will evaluate the safety and antitumor effects of abiraterone tablet formulation administered with a low dose glucocorticoid in a fasted state for up to 12 months for each stage. As of Protocol Amendment 4, all patients who have completed 12 cycles of abiraterone acetate treatment and continue to receive clinical benefit from such a treatment will enter Stage 4 and receive abiraterone acetate in a fasted condition with a low-dose glucocorticoid. Patients will continue in Stage 4 for an additional 24 cycles. After patients complete the last study visit, they will be followed every 3 months for disease progression and survival for up to 3 years. Serial pharmacokinetic samples will be collected during Stages 1 and 2. Efficacy and safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Men with histologically, cytologically, or biochemically confirmed adenocarcinoma of the prostate
* On-going androgen deprivation with serum testosterone <50 ng/dL (<2.0nmol/L)
* Serum potassium >=3.5 mmol/L
* Eastern Cooperative Oncology Group (ECOG) Performance Status score <2 (Karnofsky Performance Status >=50%)
* No history of adrenal insufficiency or hyperaldosteronism
* Any acute toxicities of prior chemotherapy, radiotherapy have resolved to a NCI CTCAE (version 3.0) grade of <=1 (chemotherapy induced alopecia and grade 2 neuropathy are excluded from this consideration)
* No radiotherapy, chemotherapy, or immunotherapy within 30 days of administration of the study drug 1 (SD1) on Day 1
* No surgery or local prostatic intervention within 28 days of the first dose (any clinically relevant sequelae from the surgery must have resolved prior to SD1 on Day 1)
* Agrees to protocol-defined use of effective contraception
* Life expectancy >12 weeks

Exclusion Criteria:

* Active or uncontrolled autoimmune disease that may require corticosteroid therapy
* Serious or uncontrolled co-existent non-malignant disease, including active and uncontrolled infection
* Uncontrolled hypertension
* Protocol-defined laboratory values
* Clinically significant heart disease as evidenced by a myocardial infarction in the past 12 months, severe or unstable angina, or New York Heart Association (NYHA) Class III or IV heart disease (patients with a history of atherosclerotic vascular disease requiring coronary or peripheral artery bypass surgery may be enrolled provided the surgery occurred at least 2 years prior to enrollment and after consultation with a cardiologist to insure that the disease is stable)
* Other malignancy within the previous 5-years other than basal cell or squamous cell carcinomas of skin with a >30% probability of recurrence within 12 months
* History of gastrointestinal disorders (medical disorders or extensive surgery) which may interfere with the absorption of the study medication
* Condition or situation which, in the investigator's opinion, may put the patient at significant risk, may confound the study results, or may interfere significantly with patient's participation in the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2007-07; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Mean plasma concentrations of abiraterone | Stage 1 predose Day 1, Days 2-4, Days 8-11; Stage 2 Day 1 Cycles 4, 7, 10
Maximum plasma concentrations of abiraterone | Stage 1 predose Day 1, Days 2-4, Days 8-11; Stage 2 Day 1 Cycles 4, 7, 10
Time to reach the maximum plasma concentration of abiraterone | Stage 1 predose Day 1, Days 2-4, Days 8-11; Stage 2 Day 1 Cycles 4, 7, 10
Area under the plasma-concentration-time curve from time 0 to the last quantifiable concentration of abiraterone | Stage 1 predose Day 1, Days 2-4, Days 8-11; Stage 2 Day 1 Cycles 4, 7, 10
Area under the plasma-concentration-time curve from time 0 to infinite time of abiraterone | Stage 1 predose Day 1, Days 2-4, Days 8-11; Stage 2 Day 1 Cycles 4, 7, 10
Elimination half-life of abiraterone | Stage 1 predose Day 1, Days 2-4, Days 8-11; Stage 2 Day 1 Cycles 4, 7, 10
Steady state trough concentration of abiraterone | Stage 1 predose Day 1, Days 2-4, Days 8-11; Stage 2 Day 1 Cycles 4, 7, 10

SECONDARY OUTCOMES:
Number of participants affected by an adverse event | Up to 30 days after the last dose of study medication
Number of patients with serum prostate specific antigen (PSA) decline according to PSA Working Group criteria | Screening; Stage 1 Day 14; Stages 2-3 Day 1, Cycles 1-12; Stage 4 every 3 cycles past Cycle 12
Number of patients with circulating tumor cells isolated from peripheral blood samples defined by cell counts | Screening; Stage 1 Days 1 and 8; Stage 2 Day 1 Cycless 1, 4, 7, and 10; Stage 4 every 3 cycles past Cycle 12
Number of patients with circulating tumor cells isolated from peripheral blood samples defined by molecular characterization | Screening; Stage 2 Day 1 Cycle 1

CONTACTS AND LOCATIONS:
Overall Officials: Cougar Biotechnology Clinical Trial, Study Director — Cougar Biotechnology, Inc.
Locations (3):
- Los Angeles, California, United States
- United Kingdom (2):
  - Glasgow
  - Sutton

REFERENCES:
- See also: A Pharmacokinetics Study to Assess the Oral Administration of CB7630 (Abiraterone Acetate) Capsule Formulation and Tablet Formulation in Patients with Prostate Cancer — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=2394&filename=CR016933_CSR.pdf